CLINICAL TRIAL: NCT03499873
Title: A Randomized, Multicenter, Double Masked, Placebo Controlled, Parallel Group, Bioequivalence Study to Evaluate the Clinical Equivalence and Safety of Nepafenac 0.3% Ophthalmic Suspension (Manufactured by Indoco Remedies Ltd. for Actavis LLC) With IlevroTM (Nepafenac Ophthalmic Suspension), 0.3% of Alcon Laboratories, Inc. for the Treatment of Pain and Inflammation Associated With Cataract Surgery.
Brief Title: Clinical Endpoint Study of Nepafenac 0.3% Opthalmic Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCTM/NEPA/2017
Record Dates: First submitted 2018-03-23; First posted 2018-04-17 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nepafenac 0.3% Opthalmic Suspension (Experimental): Test product manufactured by Indoco Remedies, Ltd for Actavis LLC.
  Interventions: Drug: Nepafenac 0.3% Oph Susp
- Ilevro 0.3% Opthalmic Suspension (Active Comparator): Reference product manufactured by Alcon Laboratories Inc.
  Interventions: Drug: Nepafenac 0.3% Oph Susp (reference)
- Placebo (vehicle) Opthalmic Suspension (Placebo Comparator): Placebo (vehicle) manufactured by Indoco Remedies, Ltd for Actavis LLC.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Nepafenac 0.3% Oph Susp — Nepafenac 0.3% Ophthalmic suspension (experimental product)
  Arms: Nepafenac 0.3% Opthalmic Suspension
Drug: Placebos — Placebo
  Arms: Placebo (vehicle) Opthalmic Suspension
Drug: Nepafenac 0.3% Oph Susp (reference) — Nepafenac 0.3% Ophthalmic suspension (Innovator)
  Arms: Ilevro 0.3% Opthalmic Suspension

SUMMARY:
A randomized, multicenter, double masked, placebo controlled, parallel group, bioequivalence study to evaluate the clinical equivalence and safety of Nepafenac 0.3% ophthalmic suspension (manufactured by Indoco remedies Ltd. for Actavis LLC) with IlevroTM (Nepafenac ophthalmic suspension), 0.3% of Alcon Laboratories, Inc. for the treatment of pain and inflammation associated with cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females, 18 years of age or older who have a cataract and are expected to undergo cataract extraction.
2. No aqueous cells, no visible aqueous flare and no significant ocular pain in the selected eye noted during the Screening visit by slit-lamp examination.
3. Study subjects must have provided IRB approved written informed consent using the latest version of the IRB informed consent form. In addition, study subjects must sign a HIPAA authorization, if applicable.
4. Study subjects should be literate and willing to complete the subject diary regularly as directed.
5. Study subjects must be in good health and free from any clinically significant disease apart from indication under study.
6. Females of child bearing potential (WOCBP*) must not be pregnant or lactating at baseline visit (as documented by a negative urine pregnancy test with a minimum sensitivity of 25 IU/L or equivalent units of beta-human chorionic gonadotropin (Beta-HCG) at screening and urine pregnancy at baseline.
7. Female subjects of childbearing potential must be willing to use an acceptable form of birth control from the day of the first dose administration to 30 days after the last administration of IP. For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (Medroxyprogesterone acetate-stabilized for at least 3 months); vaginal contraceptive; contraceptive implant; double barrier methods (e.g. condom and spermicide); Nuvaring vaginal hormonal birth control, IUD, or abstinence with a second method of birth control should the subject become sexually active. A sterile sexual partner is NOT considered an adequate form of birth control.
8. All male subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration (to 30 days after the last administration of study drug). Please see acceptable forms for "Female" birth control above. Abstinence is an acceptable method of birth control for males.
9. Study subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required scheduled study visits.
10. Study subjects must be willing to refrain from using any other treatments other than the investigational product.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy during the course of the study and for 30 days after last study dose.
2. Females of childbearing potential who do not agree to utilize an adequate form of contraception.
3. Current or past history of severe hepatic or renal impairment, uncontrolled diabetes mellitus, rheumatoid arthritis or bleeding tendencies.
4. Current or history within two months prior to baseline of clinically significant ocular disease, e.g., corneal denervation, corneal epithelial defects, severe dry eye syndrome, ocular trauma to the operative eye, corneal edema, proliferative diabetic retinopathy in the operative eye or ocular infection.
5. In the operative eye, history of chronic or recurrent inflammatory disease, e.g., iritis, scleritis, uveitis, iridocyclitis or rubeosis iritis, lens pseudoexfoliation syndrome with glaucoma or zonular compromise.
6. Congenital ocular anomaly, e.g., aniridia or congenital cataract.
7. Iris atrophy in the operative eye.
8. Current corneal abnormalities that would prevent accurate IOP readings with the Goldmann applanation tonometer.
9. Nonfunctional nonoperative eye (visual acuity of 20/200 or worse Snellen or ETDRS).
10. Known hypersensitivity to any component of nepafenac therapy or to other nonsteroidal anti-inflammatory drug (NSAID).
11. Use within one week prior to baseline of: 1) contact lens, or 2) topical, ophthalmic or systemic NSAID.
12. Use within two weeks prior to baseline of: 1) topical ophthalmic corticosteroid, 2) topical corticosteroid, or 3) medications which may prolong bleeding time (per investigator discretion and primary care physician approval to discontinue use for surgery).
13. Use within one month prior to baseline of: 1) systemic corticosteroid, 2) high-dose salicylate therapy, or 3) topical ophthalmic prostaglandin analogs, e.g., bimatoprost, latanoprost or travoprost.
14. Use within six months prior to baseline of intravitreal or subtenon injection of ophthalmic corticosteroid.
15. Underwent within six months prior to baseline any complicated intraocular surgery or repeat ocular surgeries (e.g., cataract surgery).
16. Underwent within twelve months prior to baseline: refractive surgery, filtering surgery or laser surgery for IOP reduction.
17. History or presence of significant alcoholism or drug abuse in the past one year.
18. History or presence of significant smoking (more than 20 cigarettes or any other equivalent tobacco product/day).
19. History of hematologic disorders other than mild anemia.
20. Severe, unstable, or uncontrolled cardiovascular or pulmonary disease.
21. Therapy with an investigational agent within the past 30 days prior to screening.
22. Clinically significant hematologic and / or biochemical abnormalities based on laboratory testing.
23. Subjects who are in the investigator's best judgment at risk of visual field or visual acuity worsening as a consequence of participation in trial.
24. Use of any prescribed medication during last two weeks or OTC medicinal products during the last one week preceding the first dosing that results in drug-drug interaction with the study drug.
25. Major illness, as per investigator discretion, during 3 months before screening.
26. Subjects who are employees of site or CRO or sponsor or immediate family of employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Key-Whitman Eye Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nepafenac 0.3% Opthalmic Suspension | Ilevro 0.3% Opthalmic Suspension | Placebo (Vehicle) Opthalmic Suspension
Started | 183 | 182 | 83
Safety Population | 175 | 174 | 80
Per-Protocol Population | 144 | 143 | 58
Modified-Intent-to-Treat | 170 | 168 | 77
Completed | 163 | 162 | 56
Not Completed | 20 | 20 | 27
Not completed — Withdrawal by Subject | 4 | 6 | 1
Not completed — Subjects condition worsened | 0 | 3 | 11
Not completed — Adverse Event | 8 | 3 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Administrative reasons | 0 | 1 | 0
Not completed — Concomitant therapy | 5 | 4 | 7
Not completed — Miscellaneous | 1 | 2 | 2
Not completed — Investigational Product (IP) Missed dose compliance | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics provided for Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac 0.3% Opthalmic Suspension | Ilevro 0.3% Opthalmic Suspension | Placebo (Vehicle) Opthalmic Suspension | Total
Number analyzed (Participants) | 175 | 174 | 80 | 429
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.73) | 68.5 (9.12) | 67.0 (10.19) | 68.1 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 89 | 47 | 249
  Male | 62 | 85 | 33 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 42 | 21 | 113
  Not Hispanic or Latino | 117 | 120 | 52 | 289
  Unknown or Not Reported | 8 | 12 | 7 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 8 | 3 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 24 | 24 | 13 | 61
  White | 117 | 122 | 56 | 295
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 22 | 23 | 8 | 53
Iris Colour [Count of Participants; unit: Participants]
  Blue | 38 | 47 | 13 | 98
  Green | 8 | 11 | 9 | 28
  Grey | 2 | 1 | 2 | 5
  Hazel | 19 | 21 | 9 | 49
  Brown | 97 | 81 | 41 | 219
  Black | 11 | 13 | 6 | 30
Baseline Ocular Pain Grade in Study Eye [Count of Participants; unit: Participants] — Grade 0-5 a positive sensation of the eye, including foreign body sensation, stabbing, throbbing or aching. The scoring indicates from less severe at 0 to very severe as the grading increases.
  Participants
    Grade 0 (less severe) | 172 | 172 | 80 | 424
    Grade 1 | 1 | 1 | 0 | 2
    Grade 2 | 0 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0
    Grade 5 (most severe) | 0 | 0 | 0 | 0
    Missing | 2 | 1 | 0 | 3
Baseline Aqueous Cells Grade in Study Eye [Count of Participants; unit: Participants] — Grade 0-4 using a narrow-slit beam (0.5 mm width at least 8 mm length) at maximum luminance.
  Participants
    Grade 0 (least severe) | 173 | 173 | 80 | 426
    Grade 1 | 0 | 0 | 0 | 0
    Grade 2 | 0 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0 | 0
    Grade 4 (most severe) | 0 | 0 | 0 | 0
    Missing | 2 | 1 | 0 | 3
Baseline Aqueous Flare Grade in Study Eye [Count of Participants; unit: Participants] — Grade 0-3 using a narrow-slit beam (0.5 mm width at least 8 mm length) at maximum luminance.
  Participants
    Grade 0 (least severe) | 173 | 173 | 80 | 426
    Grade 1 | 0 | 0 | 0 | 0
    Grade 2 | 0 | 0 | 0 | 0
    Grade 3 (most severe) | 0 | 0 | 0 | 0
    Missing | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cure at Day 14
Description: Number of participants that achieved cure at Day 14 defined as a score of 0 for aqueous cells (Grade 0-4 using a narrow-slit beam (0.5 mm width at least 8 mm length) at maximum luminance), a score of 0 for aqueous flare (Grade 0-3 using a narrow-slit beam (0.5 mm width at least 8 mm length) at maximum luminance) and a score of no more than 3 for pain (Grade 0-5 a positive sensation of the eye, including foreign body sensation, stabbing, throbbing or aching). The scoring indicates from less severe at 0 to very severe as the grading increases.
Time Frame: 14 days
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Nepafenac 0.3% Opthalmic Suspension | Ilevro 0.3% Opthalmic Suspension | Placebo (Vehicle) Opthalmic Suspension
Number analyzed (Participants) | 144 | 143 | 58
Participants
  Cure | 94 | 97 | 24
  Failure | 50 | 46 | 34
Statistical Analysis 1: Comparison: Nepafenac 0.3% Opthalmic Suspension vs Ilevro 0.3% Opthalmic Suspension; Test type: Equivalence — 90% CI on the Test-to-Reference difference for the proportion of subjects with cure should be contained within the interval [-0.20, +0.20]; Mean Difference (Net) = -0.026, 90% CI 2-sided [-0.124 to 0.073]
Statistical Analysis 2: Comparison: Nepafenac 0.3% Opthalmic Suspension vs Placebo (Vehicle) Opthalmic Suspension; Test type: Superiority; p = 0.0005, ANOVA
Statistical Analysis 3: Comparison: Ilevro 0.3% Opthalmic Suspension vs Placebo (Vehicle) Opthalmic Suspension; Test type: Superiority; p = 0.0003, ANOVA

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Nepafenac 0.3% Opthalmic Suspension | Ilevro 0.3% Opthalmic Suspension | Placebo (Vehicle) Opthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/174 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/174 | 0/80
Other Adverse Events (participants affected / at risk) | 54/175 | 42/174 | 26/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nepafenac 0.3% Opthalmic Suspension (N=175) | Ilevro 0.3% Opthalmic Suspension (N=174) | Placebo (Vehicle) Opthalmic Suspension (N=80)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Altered visual depth perception (Eye disorders) | 0 | 0 | 1
Anterior chamber cell (Eye disorders) | 0 | 0 | 1
Anterior chamber disorder (Eye disorders) | 1 | 0 | 0
Anterior chamber fibrin (Eye disorders) | 1 | 0 | 0
Anterior chamber inflammation (Eye disorders) | 4 | 2 | 2
Blepharitis (Eye disorders) | 1 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Conjunctival cyst (Eye disorders) | 2 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 2 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0
Corneal oedema (Eye disorders) | 2 | 2 | 4
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 2
Eye pain (Eye disorders) | 4 | 3 | 4
Eye pruritus (Eye disorders) | 1 | 0 | 0
Eyelid exfoliation (Eye disorders) | 1 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0
Hypotony of eye (Eye disorders) | 0 | 1 | 1
Keratic precipitates (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 2 | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 3
Ocular hypertention (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 1 | 3
Photopsia (Eye disorders) | 0 | 1 | 0
Posterior capsule opacification (Eye disorders) | 4 | 1 | 2
Posterior capsule rupture (Eye disorders) | 0 | 3 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Vitreous degeneration (Eye disorders) | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Sensation of foreign body (General disorders) | 1 | 2 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibrin deposition on lens postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iris injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 2 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 1
Blood glucose increased (Investigations) | 5 | 6 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 8 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 8 | 8 | 8
Migraine (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03499873/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03499873/SAP_001.pdf